CLINICAL TRIAL: NCT04438967
Title: Brain Health in the Time of COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Miro Health (Other)
Collaborators: Johns Hopkins University (Other); University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: MIRO_001_2020
Record Dates: First submitted 2020-06-15; First posted 2020-06-19 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Brain Health
Keywords: COVID-19; neurocognitive; stroke; nervous system
MeSH Terms: conditions — COVID-19; Stroke; Neurologic Manifestations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a nationwide research program to study the neurological effects of COVID-19. It is open to the public. Healthy individuals and individuals who are or have been infected with COVID-19 are encouraged to join the effort. The study can be done at home with internet access and an iPad or iPhone. Participation takes about one hour.

To learn more, go to https://www.mirohealth.com/consent/

DETAILED DESCRIPTION:
Neurological complications have been reported in patients with COVID-19. To better understand neurological complications, a group of research hospitals are collaborating to track neurological outcomes. We know that COVID-19 can invade our nervous system, but little is known about the range of effects that COVID-19 might have on the brain. This study aims to gain real-time information about the neurological health of the U.S. population to advance knowledge of COVID-19.

At the conclusion of the study, you will receive non-medical information on your brain function as well as study findings and publications made possible by your participation. With your permission, Miro Health can also release the results of your assessment to your physician. In order for Miro Health to do this, you will be required to confirm your identity online, sign a HIPAA agreement to share the information with your physician, and to enter your physician's name, email, and contact information. Study duration will depend on the development of the COVID-19 pandemic.

To participate, you must submit a valid email. No other personally identifiable information will be gathered at this time.

To participate, you will:

Answer online questions Answer a few questions about your health Download the Miro Health app from the iTunes store Open the app and complete Miro's interactive tasks (30 mins)

Advisory: Should you feel that you have symptoms related to COVID-19, contact your healthcare provider or local community health office. Miro Health cannot provide healthcare assistance.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Access to an iPad bought in 2013 or later
* Access to stable Wi-Fi
* Access to iTunes

Exclusion Criteria for healthy:

* Below age 18
* Preexisting neurological, psychiatric, or developmental disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population is open to anyone over the age of 18 who can consent for themself.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-06-16 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Test the hypothesis that COVID-19 infection will lead to increased risk of neurological impairment | ~1 year
  Each participant's Risk Score of mild cognitive impairment will be calculated using machine learning methods on a percent range of 0-100%. Miro Mobile Assessments will measure each individual's functional performance in neurocognitive, neurobehavioral, motor, and emotional domains. Miro Mobile is a clinically-validated iPad application in use by Johns Hopkins and other research centers. Miro Questionnaires will gather each individual's demographic data. To learn more, go to https://www.mirohealth.com/consent/
  Miro Functional Assessments evaluate:
  Attention Executive function Learning and Memory Motor function Processing speed Speech and language Visuospatial function
Determine cognitive and behavioral functional patterns that predict susceptibility to neurological impairment due to COVID-19 | ~1 year
  Miro Questionnaires will gather each individual's demographic and medical history data. Miro Mobile Assessments will measure each individual's CNS functional performance.
  From this data, Miro will test the hypothesis that health indicators exist that can predict the likelihood of a COVID-19 infection leading to neurological impairment.
  Miro Functional Assessments evaluate:
  Attention Executive function Learning and Memory Motor function Processing speed Speech and language Visuospatial function

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Belfor, PhD, Principal Investigator — Miro Health; Leah Rubin, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Miro Health, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: Asadi-Pooya & Simani 2020; Leonardi et al., 2020, Wu et al., 2020 — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7151535/